CLINICAL TRIAL: NCT00942045
Title: Osteocel® Plus in Anterior Cervical Discectomy and Fusion (ACDF): Evaluation of Radiographic and Patient Outcomes
Brief Title: Osteocel® Plus in Anterior Cervical Discectomy and Fusion (ACDF)
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.OC.0802
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease in Cervical Spine
Keywords: cervical spine; ACDF; biologics; fusion rates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Biologic - Osteocel Plus — Osteocel Plus

SUMMARY:
This is a prospective, non-randomized multi-center study to compare the use of Osteocel Plus in subjects who receive ACDF surgery at one or two levels. These subjects will present with degenerative conditions in the cervical spine that are amenable to surgical treatment and will be screened prior to study enrollment. Subjects will receive Osteocel Plus, without any other biologic product, during their ACDF operation. The ACDF procedure will be conducted with a radiolucent graft containment device such that progression of fusion can be adequately assessed via radiograph. Subjects will be followed for 24-months following surgery to determine the number of study subjects that are solidly fused at or before 24 months postoperatively, and to determine the mean time to fusion. This data will be compared to published and/or retrospective data for autograft, synthetic ceramics and Bone Morphogenetic Protein (BMP).

DETAILED DESCRIPTION:
A total of 175 subjects will be selected for enrollment in this study from multiple centers. The subjects will have degenerative conditions in the cervical spine and will be undergoing ACDF surgery as treatment at one or two levels. The following eligibility criteria are designed to select subjects for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether this protocol is suitable for a particular subject.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent neck and/or arm pain unresponsive to conservative treatment for at least 6 weeks, unless clinically indicated sooner
2. Indicated for anterior fusion at one or two contiguous cervical levels (C3 to T1)
3. Objective evidence of primary diagnosis must be confirmed by appropriate imaging studies
4. 18-70 years of age at the date of written informed consent
5. Able to undergo surgery based on physical exam, medical history and surgeon judgment
6. Expected to survive at least 2 years beyond surgery
7. Willing and able to return for post-treatment exams according to the follow-up called for in the protocol
8. Signed and dated Informed Consent Form

Exclusion Criteria:

1. Patient has a mental or physical condition that would limit the ability to comply with study requirements
2. Cervical spine abnormality requiring treatment at more than two levels
3. Systemic or local infection; active or latent
4. Previous failed fusion at the operative level
5. Diseases that significantly inhibit bone healing (osteoporosis, metabolic bone disease, uncontrolled diabetes, dialysis dependent renal failure, symptomatic liver disease)
6. Undergoing chemotherapy or radiation treatment, or chronic use of steroids (defined as more than 6 weeks of steroid use within 12 months of surgery, other than episodic use or inhaled corticosteroids)
7. Pregnant, or plans to become pregnant during the study
8. Subject is a prisoner
9. Involvement in active litigation relating to the spine (worker's compensation claim is allowed if it is not contended)
10. A significant general illness (e.g., HIV, active metastatic cancer of any type) is present; subject is immunocompromised or is being treated with immunosuppressive agents that decrease the probability of survival to the two-year endpoint of the study
11. Participating in another clinical study at any time during the study participation that would confound study data

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2009-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the fusion rates of Osteocel Plus in one or two level(s) for ACDF subjects. | from pre-op to 24-month follow-up

SECONDARY OUTCOMES:
To evaluate the rate of complications for Osteocel Plus and compare to published and/or retrospective data for autograft or bone morphogenetic protein (BMP). | from pre-op to 24-month follow-up
To evaluate and compare radiographic outcome with respect to clinical outcome (function and pain). | from pre-op to 24-month post-op
To evaluate and compare each outcome with respect to surgical time and blood loss. | from pre-op to 24-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Howell, MS, Study Director — NuVasive
Locations (17):
- United States (17):
  - Shiley Center for Orthopaedic, Scripps Green Hospital, La Jolla, California
  - Stanford University, Redwood City, California
  - UCSD Department of Orthpaedic Surgery, UCSD Medical Center, San Diego, California
  - The Spine Institute, St. John's Health Center, Santa Monica, California
  - University of South Florida Department of Neurosurgery, Tampa General Hospital, Tampa, Florida
  - Pinnacle Orthopaedics, Wellstone Kennestone Hospital, Marietta, Georgia
  - Hinsdale Orthopaedic Associates, Provena Saint Joseph Medical Center, Joliet, Illinois
  - Indiana Center for NeuroSurgery, Indiana Surgery Center East, Indianopolis, Indiana
  - Columbia Orthopaedic Group, Boone Hospital Center, Columbia, Missouri
  - NWREI (for Ortho Montana), Billings, Montana
  - Buffalo Spine Surgery, Kenmore Mercy, Lockport, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Center for Advanced Orthopaedics, Adena Bone and Joint Center, Chillicothe, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Spine Team Texas, Texas Health Harris Methodist Hospital Southlake, Southlake, Texas
  - Winchester Medical Center, Winchester, Virginia
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- See also: NuVasive, Inc. — http://www.nuvasive.com